CLINICAL TRIAL: NCT03277209
Title: To Assess the Safety of Continuous IV Administration of the CXCR4 Antagonist, Plerixafor at Potentially Active Plasma Concentrations and Assess Its Impact on the Immune Microenvironment in Patients With Advanced Pancreatic, High Grade Serous Ovarian and Colorectal Adenocarcinomas
Brief Title: To Assess the Safety of Continuous IV Administration of Plerixafor and Assess Impact on the Immune Microenvironment in Patients With Pancreatic, Ovarian and Colorectal Adenocarcinomas
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: terminated due to slow accrual
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1508016466
Record Dates: First submitted 2017-09-06; First posted 2017-09-08 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- All Subjects (Experimental): Plerixafor will be administered via IV as a continuous 7 day intravenous infusion starting at a dose of 20 ug/kg/hr and subsequent dose levels of 40, 80 and 120 ug/kg/hr
  Interventions: Drug: Plerixafor

INTERVENTIONS:
Drug: Plerixafor — Plerixafor will be administered via IV as a continuous 7 day intravenous infusion starting at a dose of 20 ug/kg/hr and subsequent dose levels of 40, 80 and 120 ug/kg/hr

SUMMARY:
A dose escalation trial to assess the safety of plerixafor in patients with advanced pancreatic, high grade serous ovarian and colorectal cancer. To identify the proof of mechanism, by demonstrating alterations in T-cell tumour distribution, ideally associated with loss of tumour cells, measured by immunostaining, and changes in FDG uptake.

DETAILED DESCRIPTION:
This is a prospective, non-randomised, open label, Phase I, dose escalation trial of plerixafor in patients with histological documentation of advanced pancreatic, high grade serous ovarian or colorectal adenocarcinoma. We will investigate the feasibility of administering plerixafor in terms of safety, and will try to identify the proof of mechanism in patients. This trial will follow the standard 3+3, Phase I trial design, leading to a treatment expansion phase to confirm the RP2D.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16 years or over (In the US, aged 18 years or over only).
* Dose escalation phase only: Patients with inoperable, histologically proven locally advanced or metastatic pancreatic, high grade serous ovarian or colorectal adenocarcinoma, refractory to conventional chemotherapy or a patient who has declined conventional chemotherapy OR;
* Treatment expansion phase only: Patients with inoperable, histologically proven locally advanced or metastatic pancreatic, refractory to conventional chemotherapy or a patient who has declined conventional chemotherapy.
* Tumour lesions considered to be accessible for core biopsy and immunostaining assessment.
* ECOG performance status 0-1.
* Life expectancy of at least 12 weeks.
* All women of child-bearing potential and all sexually active male patients must agree to use effective contraception methods throughout the trial and for 3 months after the final dose of trial drug.

Exclusion Criteria:

* Inadequate haematological function defined by:

  * Absolute neutrophil count (ANC) <1.5 x 109/L
  * Absolute lymphocyte count <1.0 x 109/L (counts shall be rounded to the nearest tenth. (e.g. 0.96 will be rounded to 1.0 x 109/L))
  * Haemoglobin <9.0 g/dL (90 g/L) (may be increased to this level with transfusion as long as there is no evidence of active bleeding)
  * Platelets <100 x 109/L
  * Clotting; INR >1.3
* Inadequate renal function defined by calculated creatinine clearance by Cockcroft-Gault of <50 ml/min.
* Inadequate hepatic function defined by:

  * Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) >2.5 x upper limit of normal (ULN) or >5 x in the presence of liver metastases
  * Total bilirubin >1.5 x ULN
* Current treatment (within 28 days of entry) with chemotherapy, steroids or other immunosuppressive drugs.
* Significant acute or chronic medical or psychiatric condition, disease or laboratory abnormality which in the judgment of the Investigator would place the patient at undue risk or interfere with the trial.
* Cardiac co-morbidity:

  * Past history of significant rhythm disturbance (e.g. SVT, AF or ventricular irregularities)
  * Requirement for pacemaker
  * Myocardial infarction in the previous 6 months
  * Known medical history of proven postural hypotension.
* Active infection.
* Patients with known allergy to plerixafor or its excipients.
* Patients known to have hepatitis B, hepatitis C or HIV infection.
* Participation in any other interventional clinical trial
* Women, who are pregnant, plan to become pregnant or are lactating (during the trial or for up to 3 months after the last dose)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Causality of adverse events (AEs) and serious adverse events (SAEs) and grading according to NCI CTCAE v.4.03. | From baseline through Day 56
  Assess safety of continuous IV administration of plerixafor in doses needed to achieve and maintain circulating levels similar to those active in a murine model of PDAC (2 μg/ml)

SECONDARY OUTCOMES:
Assessment of metabolic changes in tumour using non-invasive imaging (18FDG-PET) | From baseline through Day 56
  To explore objective anticancer clinical impact of this strategy.

OTHER OUTCOMES:
Change in T cell distribution within tumour regions within primary or metastatic lesions (e.g. CD3+ T cell accumulation in cancer cell "nests") | From baseline through Day 56
  To explore relationships between intratumoural T-cell distribution, CXCR4 and CXCL12 immunostaining and other potential biomarkers of immune activation in tissue and blood, such as circulating CD34+ cell counts and diurnal cortisol variation.
Changes in circulating tumour ctDNA levels within plasma, during and after treatment. | From baseline through Day 56
Changes in proliferation and apoptosis markers (e.g. Ki67/Mib1), changes in tumour cell populations in samples. | From baseline through Day 56
  To assess modulation of the immune tumour microenvironment following CXCR4 inhibition by plerixafor administration.
Changes in immune cytokine serum levels. | From baseline through Day 56
T cell receptor (TCR) sequencing in tumour tissue. | From baseline through Day 56
DNA and RNA sequencing in tumour tissue. | From baseline through Day 56
Evidence of systemic pharmacodynamic response to CXCR4i, such as increase in CD34+ cell numbers in blood. | From baseline through Day 56
Correlation between changes in T cell distribution and diurnal cortisol variation. | From baseline through Day 56

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeta Popa, MD, Principal Investigator — Weill Medical College of Cornell University; Duncan Jodrell, MD, Study Chair — Cambridge University Hospitals NHS Foundation Trust
Locations (2):
- Weill Cornell Medical College, New York, New York, United States
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, United Kingdom